CLINICAL TRIAL: NCT03456544
Title: Vancomycin-Associated Acute Kidney Injury: A Cross-Sectional Study From a Multi- Center in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Cui Yimin, Chief pharmacist, Peking University First Hospital
Other Study IDs: 20180122
Record Dates: First submitted 2018-02-01; First posted 2018-03-07 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Vancomycin; Staphylococcal Infections; Adverse Effect; Acute Kidney Injury; Cross-sectional Study
MeSH Terms: conditions — Staphylococcal Infections; Acute Kidney Injury | interventions — Vancomycin

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- VAN-AKI: Patients who had vancomycin associated acute kidney injury.
  Interventions: Drug: Vancomycin
- None VAN-AKI: Patients who didn't have vancomycin associated acute kidney injury.

INTERVENTIONS:
Drug: Vancomycin — Patients who have vancomycin associated acute kidney injury will be in the Van-AKI group, and those who don't have vancomycin associated acute kidney injury will be in the none VAN-AKI group.
  Groups: VAN-AKI

SUMMARY:
The objective of this study was to investigate the current situation of vancomycin (VAN)-associated acute kidney injury (VA-AKI) in China and identify the risk factors for VA-AKI, as well as to comprehensively examine the risk related to concurrent drug use. Further, the investigators assessed the outcomes of patients who developed VA-AKI and the risk factors for these outcomes. Finally, the investigators aimed to provide suggestions for improving the prevention and treatment of VA-AKI in China.

ELIGIBILITY:
Inclusion Criteria:

* Using Vancomycin
* ≥18 years old

Exclusion Criteria:

* Medical records were incomplete
* Had been diagnosed with stage 5 CKD or were regularly receiving dialysis
* SCr were not being adequately monitored to detect the development of AKI
* Had undergone nephrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who use vancomycin from all centers.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Vancomycin-associated acute kidney injury(VAN-AKI) occuration rate | 1 year

SECONDARY OUTCOMES:
VAN-AKI detection rate | 1 year
TDM detction rate | 1 year
0h Serum creatinine detction rate | 1 year
48h Serum creatinine detction rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China